CLINICAL TRIAL: NCT04317326
Title: "Mid- and Long-term Effectiveness of Positive Airway Pressure in OHS After an Acute-on-chronic Hypercapnic Respiratory Failure"
Brief Title: "Post-acute Pickwick Study" (Postacute-Pick-2020)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the "Philips alert " we could not get the treatment equipment and the public grands expired
Sponsor: Juan F. Masa (Other)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Juan F. Masa, Principal Investigator, Sociedad Española de Neumología y Cirugía Torácica
Organization: Sociedad Española de Neumología y Cirugía Torácica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI19/00955
Record Dates: First submitted 2020-02-14; First posted 2020-03-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Acute on Chronic Hypercapnic Respiratory Failure; Obesity Hypoventilation Syndrome (OHS)
Keywords: Hypercapnic respiratory failure; Obesity; Non invasive mechanical ventilation; CPAP
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Respiratory Insufficiency; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, open label, randomized controlled trial with two sequential phases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Life style modification (Experimental): "Lifestyle modifications" group (Control) will consist of a 1,000-calorie/day diet and to maintain proper sleep hygiene and habits (avoid supine decubitus position, maintain regular sleep habits and exercise, not take sedatives, stimulants, alcohol, tobacco or heavy meals within four hours before bedtime). Oxygen therapy can be prescribed by the treating team using standard criteria (awake PaO2 <55 mmHg or room air oxygen saturation below 88% (Masa JF et al. J Clin Sleep Med. 2016 ;12:1379-88)
  Interventions: Procedure: "Lifestyle modifications" group (Control)
- Life style modificacion and automatic NIV(AVAPS-AE) (Active Comparator): Automatic NIV: In addition to lifestyle modification and oxygen (if required), the ventilator will be adjusted to a range of predetermined parameters with the intelligent ventilation mode (pressure of intelligent support with guaranteed volume with automatic backup frequency) with the following adjustment: maximum pressure: 35 cmH2O; respiratory rate: automatic; maximum pressure support: 20 cm H2O; minimum pressure support: 4 cmH2O; maximum EPAP pressure: 15 cmH2O; minimum EPAP pressure: 4 cmH2O; and tidal volume (Vt) based on 8-10 ml/kg of predicted body weight. These parameters may be modified according to patient tolerance or non-compensated leak.
  Interventions: Procedure: Automatic NIV
- Life style modification and titrated NIV(S/T mode) (Experimental): In-laboratory polysomnographic NIV titration will be performed according to published guidelines (Berry R et al JCSM 2010). In addition to lifestyle modification and oxygen (if required), home NIV therapy with fixed pressures will be started. The ventilator mode will be a bilevel PAP with backup respiratory rate (BIPAP S/T mode). The ventilator adjustment will be firstly performed in awake situation and then during sleep by means of a PSG.
  Interventions: Procedure: CPAP treatment group
- Life style modification and titrated CPAP (Active Comparator): In-laboratory polysomnographic CPAP titration will be performed according to published guidelines (SEPAR guideline or AASM guideline). In addition to lifestyle modification and oxygen (if required), home CPAP therapy at a fixed pressure will be initiated.
  Interventions: Procedure: NIV treatment groups

INTERVENTIONS:
Procedure: "Lifestyle modifications" group (Control) — It will consist of a 1,000-calorie/day diet and to maintain proper sleep hygiene and habits (avoid supine decubitus position, maintain regular sleep habits and exercise, not take sedatives, stimulants, alcohol, tobacco or heavy meals within four hours before bedtime). Oxygen therapy can be prescribed by the treating team using standard criteria (awake PaO2 <55 mmHg or room air oxygen saturation below 88% (Masa JF et al. J Clin Sleep Med. 2016 ;12:1379-88). The treatment period will be three months.
  Arms: Life style modification
Procedure: Automatic NIV — In addition to lifestyle modification and oxygen (if required), the ventilator will be adjusted to a range of predetermined parameters with the intelligent ventilation mode (pressure of intelligent support with guaranteed volume with automatic backup frequency) with the following adjustment: maximum pressure: 35 cmH2O; respiratory rate: automatic; maximum pressure support: 18 cm H2O; minimum pressure support: 4 cmH2O; maximum EPAP pressure: 15 cmH2O; minimum EPAP pressure: 4 cmH2O; and tidal volume (Vt) based on 8-10 ml/kg of predicted body weight, being able to be modified according to tolerance.The treatment period will be three months.
  Arms: Life style modificacion and automatic NIV(AVAPS-AE)
Procedure: CPAP treatment group — In-laboratory polysomnographic CPAP titration will be performed according to published guidelines for CPAP titration (SEPAR guideline or AASM guideline).In addition to lifestyle modification and oxygen (if require), a home titrated CPAP therapy will be initiated.The treatment period will be three years.
  Arms: Life style modification and titrated NIV(S/T mode)
Procedure: NIV treatment groups — In-laboratory polysomnographic NIV titration will be performed according to published guidelines In addition to lifestyle modification and oxygen (if required) home NIV therapy with fixed pressures will be started. The ventilator mode will be a bilevel pressure in S/T mode. The ventilator adjustment will be firstly performed in awake situation and then during sleep by means of a PSG. The treatment period will be three years.
  Arms: Life style modification and titrated CPAP

SUMMARY:
We propose to carry out a large multicentric, multinational, randomized controlled trial with two phases (two sequential randomized controled trials) to answer two questions: 1) Should hospitalized patients with recently diagnosed OHS be discharged from the hospital on an auto-titratable NIV treatment until the diagnosis of OHS is confirmed in 3 months? 2) Is the long-term effectiveness of outpatient titrated CPAP non-inferior to titrated NIV in ambulatory patients with OHS 3 months after hospital discharge? Clinical practice, multicenter open-label controlled randomized clinical trial with preset allocation rate (1:1) with two parallel-groups conducted in centers from Spain, France, Portugal and USA. The study will have two phases with two randomizations. The first phase will be a superiority study and the second phase will be a non-inferiority study.

DETAILED DESCRIPTION:
Objectives: First phase (medium-term): To evaluate the medium-term (3 months) efficacy of automatically adjusted noninvasive ventilation (NIV) treatment versus "life style modifications" treatment in obesity hypoventilation syndrome (OHS) after an episode of acute-on-chronic hypercapnic respiratory failure. The main outcome will be a composite that includes hospital resource utilization (hospital and ICU admissions and emergency department visits for any cause) and all-cause mortality. Key secondary outcomes will include incident cardiovascular events (new hypertension diagnosis or initiation of anti-hypertensive treatment, atrial fibrillation, hospitalization for nonfatal myocardial infarction or unstable angina, percutaneous coronary interventions, nonfatal stroke or transient ischemic attack or for acute heart failure episode, and cardiovascular death), blood pressure, arterial blood gases, clinical symptoms and quality of life. Second phase (long-term): Evaluate the long-term efficacy (36 months) of manually titrated NIV treatment versus manually titrated CPAP treatment in OHS after 3 months of an episode of acute-on-chronic hypercapnic respiratory failure, with a composite outcome of hospital resource utilization (hospital and ICU admissions, emergency department visits) and all-cause mortality analyzed as the primary outcome. Incident cardiovascular events, blood pressure, arterial blood gases, clinical symptoms and quality of life will be the main secondary outcomes.

Methods: Prospective, multinational, randomized open-label controlled trial with two parallel arms: 1,110 hospitalized patients with newly diagnosed OHS with acute-on-chronic hypercapnic respiratory failure treated with invasive or noninvasive mechanical ventilation who survive hospitalization and available for hospital discharge will be randomized to either automatically adjusted NIV (555 patients) or "life style modifications" (555 patients) for three months. Subsequently, both automatically adjusted NIV and "life style modifications" arms will be re-randomized to polysomnographically adjusted CPAP or to polysomnographically adjusted NIV groups to complete 36 months of follow up. The first phase of the proposal is a superiority study and the second phase is a non-inferiority study. The primary outcome and its components will be analyzed by a mixed-effects model with negative binomial. A mixed-effects Cox model will be used for hospital resource utilization, new cardiovascular events and overall survival. Other secondary outcomes such as repeated measures derived from the arterial blood gases (i.e. PaCO2, PaO2, pH, calculated bicarbonate), blood pressure, health-related quality of life tests and Epworth Sleepiness Scale during the follow-up will be analyzed by a linear mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

1. º.- Patient between 18 and 85 years old.
2. º.- With diagnosis of OHS (according to Obesity (BMI ≥30 kg/m2) and Hypercapnic respiratory failure (PaCO2 ≥45 mmHg at hospital discharge) not secondary to other causes.
3. º - Hospitalized for an episode of acute-on-chronic hypercapnic respiratory failure, receiving hospital therapy with invasive or noninvasive ventilation, and just deemed stable for home discharge."
4. º.- No NIV or CPAP home therapy in the last 6 months[*].
5. º.- Being able to tolerate and correctly execute a 15-minute test with automatic NIV (AVAPS-AE) and another 15-minute test with fixed CPAP treatments during wakefulness.
6. º.- Providing informed consent (dated and signed).

[*] Patients who have objective evidence of minimal PAP therapy during the 6 months prior to hospital admission (i.e. average daily use of less than 2 hours of PAP therapy) can also be enrolled at the discretion of the investigators if they feel the patient is now more interested in being adherent to NIV therapy.

Inclusion criteria for the second phase of the study:

1º.- Included three months ago in the first phase of the study (followed by a washout period of 5 days).

Exclusion Criteria:

Exclusion criteria for the first phase of the study:

1. º.- With moderate or severe chronic obstructive pulmonary disease (FEV1<70% of predicted when FEV1/FVC is below 70%).
2. º.- With neuromuscular disease, thoracic wall or metabolic disease that may cause diurnal hypercapnia.
3. º.- Inability to maintain a patent airway or adequately clear secretions.
4. º.- With bullous lung disease or with pneumothorax.
5. º.- With bypassed upper airway (i.e. endotracheal tube or tracheostomy).
6. º.- With anatomical abnormalities of the craniofacial structure leading to cerebral spinal fluid leaks, abnormalities of the cribriform plate, and/or pneumocephalus.
7. º.- At risk for aspiration of gastric contents.
8. º.- Diagnosed with acute sinusitis or otitis media.
9. º.- With active hemoptysis or epistaxis if presenting a risk of causing pulmonary aspiration of blood.
10. º.- With symptomatic hypotension.
11. º.- With clinical diagnosis of narcolepsy or restless leg syndrome.
12. º.- Psycho-physical incapacity to complete questionnaires.
13. º.- With diagnosis of chronic illness that might interfere the evaluation using quality of life questionnaires (neoplasia, severe chronic pain of any type, and any other severe chronic debilitating illness).
14. º.- Suffering other clinically relevant disease that, under the opinion of the investigator, might affect the evaluations of efficacy or safety.
15. º.- Participating simultaneously in other clinical study with intervention (or without intervention at the discretion of the investigator and with the consent of the Sponsor) or had participated in other clinical study with intervention within the last 30 days before the inclusion in this study. [‡]
16. º.- If for any reason (planned surgery [including bariatric surgery], trips of long duration, etc.) would not be able to receive the treatment and/or attend the follow-up visits of this study within the next three years and three months.
17. º.- Persons deprived of liberty by judicial or administrative decision, persons under psychiatric treatment and persons placed in a health or social institution for purposes other than those of this clinical study.
18. º.- Adults who are subject to a legal protection measure or who are unable to express their consent.

[‡] This prohibition shall be maintained for the duration of the patients' participation in the study. This is because, if patients received other treatments, it could be difficult to interpret the causality of the results obtained (whether beneficial or harmful effects) and the possible contraindications.

vi. Exclusion criteria for the second phase of the study:

1º.- With apnea hypopnea index (AHI) lower than 5 (absence or very mild obstructive sleep apnea).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Medium-term composite hospital resource utilization-mortality | 3 months
  Primary (medium-term from the first phase or RCT): the medium-term efficacy of automatic NIV treatment versus "lifestyle modifications" treatment in OHS measuring as primary outcome a composite including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events
Long-term composite hospital resource utilization-mortality | 3 years
  Primary (long-term from the second phase or RCT): the long-term efficacy of titrated CPAP therapy versus titrated NIV therapy in OHS measuring as primary outcome a composite including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events

SECONDARY OUTCOMES:
Hospital admissions | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Separately the components of the primary outcome: hospital admissions measured as the number of events
ICU admissions | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Separately the components of the primary outcome: ICU admissions measured as the number of events
Emergency department visits | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Separately the components of the primary outcome: emergency department visits for any cause measured as the number of events
All-cause mortality | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Separately the components of the primary outcome: All-cause mortality number
Duration of hospital admissions | During 3 months and during 3 years for the first and second phase or sequential RCTs respectively
  Duration of hospital admissions measured in days of hospital admission
Duration of ICU admissions | During 3 months and during 3 years for the first and second phase or sequential RCTs respectively
  Duration of ICU admissions measured in days of ICU admission
Number of patients who change of the allocated arms | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients who change of the allocated arms
Causes of change of the allocated treatment | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Causes of change of the allocated arms
Clinical symptoms: lower extremity edema | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: unrefreshing sleep | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: morning fatigue | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: nocturia | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: headache | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: tiredness | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: morning confusion | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients into four levels of frequency (no, sometimes, usually and always)
Clinical symptoms: dysnea | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of patients with dysnea according to the Medical Research Council scale classified into five levels of intensity (from 0 to 4)
Clinical symptoms: sleepiness | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Level of perceived sleepiness measured by the Epworth Sleepiness Scale
Health related quality of life (HRQL): Functional Outcomes of Sleep Questionnaire-- FOSQ-- | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Scoring of Functional Outcomes of Sleep Questionnaire-- FOSQ---
Health related quality of life (HRQL): European health-related quality of life questionnaire (EuroQol) EQ-5D-5L | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Scoring of European health-related quality of life questionnaire (EuroQol) EQ-5D-5L
Health related quality of life (HRQL): Subjective state of illness on a visual analogical scale: Visual Analogical Well-being Scale -VAWS (Masa JF et al. Sleep Breath. 2011;15:549-59) (EuroQol) EQ-5D-5L | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Scoring of Subjective state of illness on a visual analogical scale: Visual Analogical Well-being Scale -VAWS (Masa JF et al. Sleep Breath. 2011;15:549-59) measured in percentage.
Arterial blood gases (ABG): PaO2 | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  PaO2 in mmHg
Arterial blood gases (ABG): PaCO2 | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  PaCO2 in mmHg
Arterial blood gases (ABG): Bicarbonate | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  bicarbonate measured in mmol/L
Arterial blood gases (ABG): pH | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  pH
Weight | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  weight in Kg
Standardized blood pressure measures | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Systolic and diastolic blood pressure measured in mmHg
Incidence of cardiovascular events: systemic hypertension | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of hypertension diagnosis or initiation of a new anti-hypertensive treatment
Incidence of cardiovascular events: arrhythmia | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of arrhythmia
Incidence of cardiovascular events: nonfatal myocardial infarction | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of nonfatal myocardial infarction
Incidence of cardiovascular events: hospitalization for unstable angina | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of hospitalization for unstable angina
Incidence of cardiovascular events: coronary percutaneous interventions | After 3 months and after 3 years for first and second phases or sequential RCTs respectively
  Incidence of coronary percutaneous interventions
Incidence of cardiovascular events: nonfatal stroke or transient ischemic attack | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Incidence of nonfatal stroke or transient ischemic attack
Incidence of cardiovascular events: heart failure episode | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of heart failure episode
Incidence of cardiovascular events: cardiovascular death | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Incidence of cardiovascular death.
Incidence of adverse event | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of adverse events according to Treatment-Related Adverse Events as assessed by CTCAE v5.0
Cost-effectiveness analysis based on the primary outcome and quality adjusted life year (QALY) | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Differences in within trial costs will be related with the differences in effectiveness (primary outcome and QALY) between arms using a probabilistic approach to calculate the cost-effectiveness plane.
Number of oro-tracheal intubation | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Number of the tracheal intubations
Duration of tracheal intubation | During 3 months and during 3 years for the first and second phases or sequential RCTs respectively
  Duration of tracheal intubation

OTHER OUTCOMES:
A composite outcome in adherent vs. non-adherent to PAP therapy subgroups | During 3 months for the first phase or RCT
  Efficacy of automatic NIV treatment versus "lifestyle modifications" treatment measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events comparing adherent vs. non-adherent to PAP therapy subgroups (lower and higher of a mean of 4 h/day)
A composite outcome in adherent vs. non-adherent to PAP therapy subgroups | During 3 years for the second phase or RCT
  Efficacy of automatic NIV treatment versus CPAP treatment measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events comparing adherent vs. non-adherent to PAP therapy subgroups (lower and higher of a mean of 4 h/days)
Subgroups according to whether hypercapnia was resolved or not | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with PaCO2 higher or lower of 45 mmHg at the end of follow-up
A composite outcome in subgroups with or without supplemental oxygen at baseline | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with or without supplemental oxygen therapy at baseline
A composite outcome in subgroups of hypercapnia severity at baseline | During 3 months and During 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with higher and lower hypercapnia at baseline (above and below of the median PaCO2 measured in mmHg)
A composite outcome in subgroups of the apnea-hypopnea index severity at baseline | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with higher and lower apnea-hypopnea index at baseline (above and below of the median apnea-hypopnea index at baseline)
A composite outcome in subgroups with or without hypertension diagnosis at baseline | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with or without hypertension diagnosis at baseline
A composite outcome in subgroups with different home care providers | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  Comparative efficacy between treatment arms measuring a composite outcome including hospital and ICU admissions, emergency department visits for any cause, and all-cause mortality measured as the number of events in the subgroups with different home care providers (i.e. AirLiquide)
Validity analysis of EQ 5D-5L test | During 3 months and during 3 years for first and second phases or sequential RCTs respectively
  To perform a validity analysis of EQ 5D-5L test

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Masa, MD, Phd, Principal Investigator — Servicio Extremeño de Salud; Babak Mokhlesi, MD, Prof, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Additional related documents such as study protocol, statistical analysis plan, and informed consent form will be available upon request from the Project principal investigator (Dr. Juan Fernando Masa). Deidentified patients' data can be requested by researchers for use in independent scientific research and will be provided following review and approval of the research proposal (including statistical analysis plan) and completion of a data sharing agreement with the Project Publications Committee. Investigator Data requests can be made anytime from 1 to 2 years after the publication of this trial. Requests should be sent to the corresponding author (Dr. Juan Fernando Masa- fmasa@separ.es).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after the publication of this tria
Access Criteria: Requests should be sent to the corresponding authors (Dr. Juan Fernando Masa- fmasa@separ.es; and Dr Babak Mokhlesi- Babak_Mokhlesi@rush.edu).

REFERENCES:
- [Background] Storre JH, Seuthe B, Fiechter R, Milioglou S, Dreher M, Sorichter S, Windisch W. Average volume-assured pressure support in obesity hypoventilation: A randomized crossover trial. Chest. 2006 Sep;130(3):815-21. doi: 10.1378/chest.130.3.815. PMID 16963680
- [Result] Masa JF, Rubio M, Findley LJ. Habitually sleepy drivers have a high frequency of automobile crashes associated with respiratory disorders during sleep. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1407-12. doi: 10.1164/ajrccm.162.4.9907019. PMID 11029353
- [Result] Teran-Santos J, Jimenez-Gomez A, Cordero-Guevara J. The association between sleep apnea and the risk of traffic accidents. Cooperative Group Burgos-Santander. N Engl J Med. 1999 Mar 18;340(11):847-51. doi: 10.1056/NEJM199903183401104. PMID 10080847
- [Result] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Result] Kessler R, Chaouat A, Schinkewitch P, Faller M, Casel S, Krieger J, Weitzenblum E. The obesity-hypoventilation syndrome revisited: a prospective study of 34 consecutive cases. Chest. 2001 Aug;120(2):369-76. doi: 10.1378/chest.120.2.369. PMID 11502631
- [Result] Masa JF, Corral J, Alonso ML, Ordax E, Troncoso MF, Gonzalez M, Lopez-Martinez S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Aizpuru F, Egea C; Spanish Sleep Network. Efficacy of Different Treatment Alternatives for Obesity Hypoventilation Syndrome. Pickwick Study. Am J Respir Crit Care Med. 2015 Jul 1;192(1):86-95. doi: 10.1164/rccm.201410-1900OC. PMID 25915102
- [Result] Castro-Anon O, Perez de Llano LA, De la Fuente Sanchez S, Golpe R, Mendez Marote L, Castro-Castro J, Gonzalez Quintela A. Obesity-hypoventilation syndrome: increased risk of death over sleep apnea syndrome. PLoS One. 2015 Feb 11;10(2):e0117808. doi: 10.1371/journal.pone.0117808. eCollection 2015. PMID 25671545
- [Result] Basoglu OK, Tasbakan MS. Comparison of clinical characteristics in patients with obesity hypoventilation syndrome and obese obstructive sleep apnea syndrome: a case-control study. Clin Respir J. 2014 Apr;8(2):167-74. doi: 10.1111/crj.12054. Epub 2013 Nov 28. PMID 24028180
- [Result] Priou P, Hamel JF, Person C, Meslier N, Racineux JL, Urban T, Gagnadoux F. Long-term outcome of noninvasive positive pressure ventilation for obesity hypoventilation syndrome. Chest. 2010 Jul;138(1):84-90. doi: 10.1378/chest.09-2472. Epub 2010 Mar 26. PMID 20348200
- [Result] Berg G, Delaive K, Manfreda J, Walld R, Kryger MH. The use of health-care resources in obesity-hypoventilation syndrome. Chest. 2001 Aug;120(2):377-83. doi: 10.1378/chest.120.2.377. PMID 11502632
- [Result] Corral J, Mogollon MV, Sanchez-Quiroga MA, Gomez de Terreros J, Romero A, Caballero C, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martinez S, de Lucas P, Marin JM, Romero O, Diaz-Cambriles T, Chiner E, Egea C, Lang RM, Mokhlesi B, Masa JF; Spanish Sleep Network. Echocardiographic changes with non-invasive ventilation and CPAP in obesity hypoventilation syndrome. Thorax. 2018 Apr;73(4):361-368. doi: 10.1136/thoraxjnl-2017-210642. Epub 2017 Nov 16. PMID 29146865
- [Result] Masa JF, Corral J, Romero A, Caballero C, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Merchan M, Egea C, Obeso A, Mokhlesi B; Spanish Sleep Network( *). Protective Cardiovascular Effect of Sleep Apnea Severity in Obesity Hypoventilation Syndrome. Chest. 2016 Jul;150(1):68-79. doi: 10.1016/j.chest.2016.02.647. Epub 2016 Feb 27. PMID 26923627
- [Result] Weitzenblum E, Kessler R, Chaouat A. [Alveolar hypoventilation in the obese: the obesity-hypoventilation syndrome]. Rev Pneumol Clin. 2002 Apr;58(2):83-90. French. PMID 12082446
- [Result] Chaouat A, Weitzenblum E, Krieger J, Sforza E, Hammad H, Oswald M, Kessler R. Prognostic value of lung function and pulmonary haemodynamics in OSA patients treated with CPAP. Eur Respir J. 1999 May;13(5):1091-6. doi: 10.1034/j.1399-3003.1999.13e25.x. PMID 10414409
- [Result] Biring MS, Lewis MI, Liu JT, Mohsenifar Z. Pulmonary physiologic changes of morbid obesity. Am J Med Sci. 1999 Nov;318(5):293-7. doi: 10.1097/00000441-199911000-00002. PMID 10555090
- [Result] Leech J, Onal E, Aronson R, Lopata M. Voluntary hyperventilation in obesity hypoventilation. Chest. 1991 Nov;100(5):1334-8. doi: 10.1378/chest.100.5.1334. PMID 1935291
- [Result] Zwillich CW, Sutton FD, Pierson DJ, Greagh EM, Weil JV. Decreased hypoxic ventilatory drive in the obesity-hypoventilation syndrome. Am J Med. 1975 Sep;59(3):343-8. doi: 10.1016/0002-9343(75)90392-7. PMID 1163544
- [Result] MacGregor MI, Block AJ, Ball WC Jr. Topics in clinical medicine: serious complications and sudden death in the Pickwickian syndrome. Johns Hopkins Med J. 1970 May;126(5):279-95. No abstract available. PMID 5419916
- [Result] Miller A, Granada M. In-hospital mortality in the Pickwickian syndrome. Am J Med. 1974 Feb;56(2):144-50. doi: 10.1016/0002-9343(74)90591-9. No abstract available. PMID 4812072
- [Result] Jennum P, Kjellberg J. Health, social and economical consequences of sleep-disordered breathing: a controlled national study. Thorax. 2011 Jul;66(7):560-6. doi: 10.1136/thx.2010.143958. Epub 2011 Jan 2. PMID 21199816
- [Result] Olson AL, Zwillich C. The obesity hypoventilation syndrome. Am J Med. 2005 Sep;118(9):948-56. doi: 10.1016/j.amjmed.2005.03.042. PMID 16164877
- [Result] Berger KI, Ayappa I, Chatr-Amontri B, Marfatia A, Sorkin IB, Rapoport DM, Goldring RM. Obesity hypoventilation syndrome as a spectrum of respiratory disturbances during sleep. Chest. 2001 Oct;120(4):1231-8. doi: 10.1378/chest.120.4.1231. PMID 11591566
- [Result] Masa JF, Corral J, Caballero C, Barrot E, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Miranda E, Mokhlesi B; Spanish Sleep Network; Garcia-Ledesma E, Sanchez-Quiroga MA, Ordax E, Gonzalez-Mangado N, Troncoso MF, Martinez-Martinez MA, Cantalejo O, Ojeda E, Carrizo SJ, Gallego B, Pallero M, Ramon MA, Diaz-de-Atauri J, Munoz-Mendez J, Senent C, Sancho-Chust JN, Ribas-Solis FJ, Romero A, Benitez JM, Sanchez-Gomez J, Golpe R, Santiago-Recuerda A, Gomez S, Bengoa M. Non-invasive ventilation in obesity hypoventilation syndrome without severe obstructive sleep apnoea. Thorax. 2016 Oct;71(10):899-906. doi: 10.1136/thoraxjnl-2016-208501. Epub 2016 Jul 12. PMID 27406165
- [Result] Masa JF, Mokhlesi B, Benitez I, Gomez de Terreros FJ, Sanchez-Quiroga MA, Romero A, Caballero-Eraso C, Teran-Santos J, Alonso-Alvarez ML, Troncoso MF, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Vazquez-Polo FJ, Negrin MA, Martel-Escobar M, Barbe F, Corral J; Spanish Sleep Network. Long-term clinical effectiveness of continuous positive airway pressure therapy versus non-invasive ventilation therapy in patients with obesity hypoventilation syndrome: a multicentre, open-label, randomised controlled trial. Lancet. 2019 Apr 27;393(10182):1721-1732. doi: 10.1016/S0140-6736(18)32978-7. Epub 2019 Mar 29. PMID 30935737
- [Result] Mokhlesi B. Obesity hypoventilation syndrome: a state-of-the-art review. Respir Care. 2010 Oct;55(10):1347-62; discussion 1363-5. PMID 20875161
- [Result] Lee WY, Mokhlesi B. Diagnosis and management of obesity hypoventilation syndrome in the ICU. Crit Care Clin. 2008 Jul;24(3):533-49, vii. doi: 10.1016/j.ccc.2008.02.003. PMID 18538199
- [Result] Berry RB, Chediak A, Brown LK, Finder J, Gozal D, Iber C, Kushida CA, Morgenthaler T, Rowley JA, Davidson-Ward SL; NPPV Titration Task Force of the American Academy of Sleep Medicine. Best clinical practices for the sleep center adjustment of noninvasive positive pressure ventilation (NPPV) in stable chronic alveolar hypoventilation syndromes. J Clin Sleep Med. 2010 Oct 15;6(5):491-509. PMID 20957853
- [Result] Mokhlesi B, Masa JF, Brozek JL, Gurubhagavatula I, Murphy PB, Piper AJ, Tulaimat A, Afshar M, Balachandran JS, Dweik RA, Grunstein RR, Hart N, Kaw R, Lorenzi-Filho G, Pamidi S, Patel BK, Patil SP, Pepin JL, Soghier I, Tamae Kakazu M, Teodorescu M. Evaluation and Management of Obesity Hypoventilation Syndrome. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2019 Aug 1;200(3):e6-e24. doi: 10.1164/rccm.201905-1071ST. PMID 31368798
- [Result] Carrillo A, Ferrer M, Gonzalez-Diaz G, Lopez-Martinez A, Llamas N, Alcazar M, Capilla L, Torres A. Noninvasive ventilation in acute hypercapnic respiratory failure caused by obesity hypoventilation syndrome and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Dec 15;186(12):1279-85. doi: 10.1164/rccm.201206-1101OC. Epub 2012 Oct 26. PMID 23103736
- [Result] Howard ME, Piper AJ, Stevens B, Holland AE, Yee BJ, Dabscheck E, Mortimer D, Burge AT, Flunt D, Buchan C, Rautela L, Sheers N, Hillman D, Berlowitz DJ. A randomised controlled trial of CPAP versus non-invasive ventilation for initial treatment of obesity hypoventilation syndrome. Thorax. 2017 May;72(5):437-444. doi: 10.1136/thoraxjnl-2016-208559. Epub 2016 Nov 15. PMID 27852952
- [Result] Murphy PB, Davidson C, Hind MD, Simonds A, Williams AJ, Hopkinson NS, Moxham J, Polkey M, Hart N. Volume targeted versus pressure support non-invasive ventilation in patients with super obesity and chronic respiratory failure: a randomised controlled trial. Thorax. 2012 Aug;67(8):727-34. doi: 10.1136/thoraxjnl-2011-201081. Epub 2012 Mar 1. PMID 22382596
- [Result] Palm A, Midgren B, Janson C, Lindberg E. Gender differences in patients starting long-term home mechanical ventilation due to obesity hypoventilation syndrome. Respir Med. 2016 Jan;110:73-8. doi: 10.1016/j.rmed.2015.11.010. Epub 2015 Nov 26. PMID 26680503
- [Result] Budweiser S, Riedl SG, Jorres RA, Heinemann F, Pfeifer M. Mortality and prognostic factors in patients with obesity-hypoventilation syndrome undergoing noninvasive ventilation. J Intern Med. 2007 Apr;261(4):375-83. doi: 10.1111/j.1365-2796.2007.01765.x. PMID 17391112
- [Result] Borel JC, Burel B, Tamisier R, Dias-Domingos S, Baguet JP, Levy P, Pepin JL. Comorbidities and mortality in hypercapnic obese under domiciliary noninvasive ventilation. PLoS One. 2013;8(1):e52006. doi: 10.1371/journal.pone.0052006. Epub 2013 Jan 16. PMID 23341888
- [Result] McArdle N, Rea C, King S, Maddison K, Ramanan D, Ketheeswaran S, Erikli L, Baker V, Armitstead J, Richards G, Singh B, Hillman D, Eastwood P. Treating Chronic Hypoventilation With Automatic Adjustable Versus Fixed EPAP Intelligent Volume-Assured Positive Airway Pressure Support (iVAPS): A Randomized Controlled Trial. Sleep. 2017 Oct 1;40(10). doi: 10.1093/sleep/zsx136. PMID 28958052